CLINICAL TRIAL: NCT07116369
Title: Enhancing Prediction of Spontaneous Bacterial Peritonitis in Liver Cirrhosis by Integrating Serum Sodium and Platelet Count With the Albumin-Bilirubin Score .
Brief Title: Prediction of SBP in Cirrhotic Patients by Platlet Count, Na and AlBl Index.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Helmy Mahmoud, Internal Medicine Resident Doctor, Sohag University
Other Study IDs: Soh-Med--25-7-10MS
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: Spontaneous bacterial peritonitis; SBP; Liver cirrhosis; ABLI score; Ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ascites patients: >18 yr old Patients with liver cirrhosis and ascites, peritoneal aspirate, ALBI score, plaltlet, serum sodium will be recorded

SUMMARY:
This study aims to evaluate whether integrating serum sodium levels and platelet count with the Albumin-Bilirubin (ALBI) score can improve the early prediction of spontaneous bacterial peritonitis (SBP) in cirrhotic patients with ascites. SBP is a common and potentially life-threatening complication of cirrhosis. Identifying at-risk patients early using simple, routine laboratory parameters could enhance risk stratification, guide monitoring strategies, and reduce associated morbidity and mortality.

Participants will be Adult patients (≥18 years) with liver cirrhosis and ascites undergoing diagnostic paracentesis at Sohag University Hospital.

DETAILED DESCRIPTION:
This is a prospective observational study designed to enhance the prediction of spontaneous bacterial peritonitis (SBP) in patients with liver cirrhosis and ascites by integrating serum sodium levels and platelet count with the Albumin-Bilirubin (ALBI) score. SBP remains a serious and potentially fatal complication in cirrhotic patients, with delayed diagnosis contributing to poor outcomes. The ALBI score, which reflects liver function objectively, along with hyponatremia and thrombocytopenia-common in cirrhosis-may provide a simple, low-cost method for early identification of patients at high risk for SBP.

The study will be conducted over 6 months at the Internal Medicine and Hepatology Units, Sohag University Hospital. All eligible adult patients (≥18 years) with liver cirrhosis and ascites who undergo diagnostic paracentesis will be screened for inclusion.

Inclusion criteria include cirrhotic patients with ascites undergoing diagnostic paracentesis.

Exclusion criteria include secondary peritonitis, advanced hepatocellular carcinoma, obstructive jaundice, recent antibiotic use (<7 days), end-stage renal disease requiring dialysis, current use of immunosuppressive therapy, and incomplete data.

Each participant will undergo clinical evaluation and laboratory testing, including serum albumin, bilirubin (for ALBI calculation), sodium, and platelet count. Ascitic fluid analysis will be performed to diagnose SBP based on PMN count ≥250 cells/mm³.

The study will assess whether a combined score (ALBI-Na-Platelet) can improve prediction accuracy. Statistical analysis will involve logistic regression and ROC curve analysis to evaluate the predictive power of the combined parameters.

All participants will provide written informed consent. The study is approved by the Medical Ethics Committee of Sohag University, Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) with liver cirrhosis and ascites who underwent diagnostic paracentesis.

Exclusion Criteria:

* obstructive jaundice
* Recent antibiotic use < 7 days
* Secondary pertonitis (bowel perforation)
* Advanced Hepatocelluar carcinoma
* End-stage renal disease requiring dialysis
* Use of immunosuppressive therapy
* Incomplete laboratory or clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (≥18 years) with liver cirrhosis and ascites who underwent diagnostic paracentesis in sohag university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of SBP, ALBI score, s.sodium, platelet count | Within 1 week
  Outcome of SBP in cirrhotic patients by measurement of ALBI score, platelet count and s.sodium

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided